CLINICAL TRIAL: NCT03055234
Title: A Phase 3, Multicenter, Randomized, Placebo-controlled Study to Evaluate Efficacy and Safety of Oral Treprostinil in Subjects With Pulmonary Hypertension Associated With Sickle Cell Disease
Brief Title: Study to Evaluate Efficacy and Safety of Oral Treprostinil in Subjects With Pulmonary Hypertension (PH) Associated With Sickle Cell Disease (SCD)
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Business decision
Sponsor: United Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TDE-SC-301
Record Dates: First submitted 2017-01-27; First posted 2017-02-16 (Actual); Last update posted 2017-04-11 (Actual); Status verified 2017-04

CONDITIONS: Pulmonary Hypertension Associated With Sickle Cell Disease
Keywords: Oral treprostinil; 6-Minute Walk Distance; PH; sickle cell
MeSH Terms: interventions — treprostinil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Oral Treprostinil (Experimental): Extended-release oral tablet for three times daily (TID) administration
  Interventions: Drug: Oral Treprostinil
- Placebo (Placebo Comparator): Placebo (sugar pill) for TID administration
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Oral Treprostinil — Extended-release oral tablet for TID administration
  Arms: Oral Treprostinil
Drug: Placebo — Matching placebo for TID administration
  Arms: Placebo

SUMMARY:
This is a multicenter, randomized (2:1; oral treprostinil:placebo), double-blind, placebo-controlled event-driven (time to pulmonary hypertension [PH] clinical worsening) study in subjects with PH associated with sickle cell disease (SCD). Once enrolled, subjects will be evaluated at Weeks 6, 12, 24, and then every 12 weeks for the duration of the study. Subjects will be permitted to enter a 48-week open-label extension period if they experience a PH clinical worsening event.

ELIGIBILITY:
Inclusion Criteria:

1. The subject must have a diagnosis of SCD confirmed by hemoglobin electrophoresis.
2. The subject has a diagnosis of symptomatic World Health Organization (WHO) Group 5.1 chronic hemolytic anemia PH.
3. The subject must have a Baseline 6MWD greater than 150 meters, in the absence of a concurrent injury, illness, or other confounding factor.
4. The subject has pulmonary function tests conducted within 6 months of Screening or during the Screening period.
5. The subject must be on stable doses of other medical therapy for at least 30 days prior to randomization with no dose adjustments, additions, or discontinuations.
6. The subject must be optimally treated with conventional PH therapy for at least 10 days prior to randomization with no additions, discontinuations, or dose changes.
7. Subjects receiving an endothelin receptor antagonist (ERA) must have been receiving therapy for greater than 90 days, and have reached and maintained a stable dose for a minimum of 30 days prior to randomization.
8. Subjects receiving calcium channel blockers must have been on a stable dose for a minimum of 3 months prior to randomization.

Exclusion Criteria:

1. The subject is pregnant or lactating.
2. The subject has previously received oral treprostinil or is receiving a phosphodiesterase type 5 inhibitor (PDE5-I).
3. The subject has received a prostacyclin within 30 days prior to start of the study, or had previous intolerance or significant lack of efficacy to any prostacyclin or prostacyclin analogue that resulted in discontinuation or inability to titrate that therapy effectively.
4. The subject has had any other background conventional therapies for PH added, removed, or doses adjusted within 10 days prior to randomization.
5. The subject has any disease associated with pulmonary arterial hypertension (PAH).
6. The subject has had a vaso-occlusive crisis, acute chest syndrome event, or unscheduled transfusion within 30 days of randomization.
7. The subject has a history of ischemic heart disease, including a previous myocardial infarction or symptomatic coronary artery disease, within 6 months prior to Screening or a left ventricular ejection fraction less than 40% assessed by either multigated angiogram (MUGA), angiography, or echocardiogram.
8. The subject has alanine aminotransferase (ALT) or aspartate aminotransferase (AST) levels 3 times or greater than the upper limit of normal, clinically significant liver disease/dysfunction, or known Child-Pugh Class B or C hepatic disease at Screening.
9. The subject has chronic renal insufficiency, as defined by the requirement for dialysis.
10. The subject has a musculoskeletal disorder, any disease that is likely to limit ambulation, or is connected to a machine that is not portable.
11. The subject has an unstable psychiatric condition or is mentally incapable of understanding the objectives, nature, or consequences of the study, or has any condition which in the Investigator's opinion would constitute an unacceptable risk to the subject's safety.
12. The subject is receiving an investigational drug, has an investigational device in place, or has participated in an investigational drug or device study within 30 days prior to Screening.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-06 (Estimated); Primary Completion 2021-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Effect of oral treprostinil compared with placebo on time to first adjudicated PH clinical worsening (morbidity or mortality) event in subjects with PH associated with SCD | Baseline until the first adjudicated PH clinical worsening event, assessed up to approximately 4 years
  Clinical worsening is defined as the occurrence of any 1 of the following events: hospitalization related to PH and/or right heart failure, initiation of an infused prostacyclin to treat worsening PH, decrease in 6-Minute Walk Distance (6MWD) >15% from Baseline directly related to disease under study.

SECONDARY OUTCOMES:
Effect of oral treprostinil compared with placebo on exercise capacity as assessed by 6-Minute Walk Distance (6MWD) | Baseline to Week 24
Effect of oral treprostinil compared with placebo on combined 6MWD/Borg dyspnea score | Baseline to Week 24
Effect of oral treprostinil compared with placebo on Borg dyspnea score | Baseline to Week 24
Effect of oral treprostinil compared with placebo on N-Terminal pro-brain natriuretic peptide (NT-proBNP) levels | Baseline to Week 24
Effect of oral treprostinil compared with placebo on maximal tricuspid regurgitant velocity (TRV) assessed by transthoracic Doppler echocardiography | Baseline to Week 24

IPD SHARING:
Plan to Share IPD: No